CLINICAL TRIAL: NCT01131455
Title: Autologous Concentrated Platelet-rich Plasma (Arthrex ACP®) for Local Application in Ankle Arthrodesis: A Prospective Outcome Analysis.
Brief Title: ACP for Local Application in Ankle Arthrodesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to the untimely death of the investigator
Sponsor: Columbia Orthopaedic Group, LLP (Other)
Responsible Party: Principal Investigator, Vicki L Jones, Sr. Research Coordinator, Columbia Orthopaedic Group, LLP
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTH-0071
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Ankle Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fusion+ACP+Autograft (Active Comparator): Standard anatomic reduction will be adhered to- neutral alignment will be employed (5° valgus, external rotation and neutral foot dorsiflexion). The arthrodesis undertaken for all groups will be the standard arthroscopic ankle arthrodesis with portals to the ankle (anterior medial / anterior lateral), skin incision only technique with dissection through the capsule and penetration to the joint. Standard debridement of the gutters, tibia osteophyte, tibia-talor joint resection and autograft preparation will be performed in the joint. Depending on randomization of the subject, (Autologous concentrated Plasma)ACP-A or ACP-DBM mixture will be added to the arthrodesis site with the joint taken through range of direct motion and reduced.
  Interventions: Biological: Autologous Concentrated Plasma
- Fusion + ACP +DBM (Active Comparator): Standard anatomic reduction will be adhered to- neutral alignment will be employed (5° valgus and external rotation and neutral foot dorsiflexion). Depending on the randomization of the subject, (Autologous Concentrated Plasma)ACP-A or ACP-DBM mixture will be added to the arthrodesis site with the joint taken through range of direct motion and then reduced.
  Interventions: Biological: Autologous Concentrated Plasma
- Standard-Fusion +Autograft only (No Intervention): Standard anatomic reduction will be adhered to- neutral alignment will be employed (5° valgus and external rotation and neutral foot dorsiflexion). The arthrodesis undertaken for all groups will be the standard arthroscopic ankle arthrodesis with portals to the ankle (anterior medial / anterior lateral), skin incision only technique with blunt dissection through the capsule and penetration to the joint. Depending on the randomization of the subject, ACP-A or ACP-DBM mixture will be added to the arthrodesis site with the joint taken through range of direct motion and then reduced.

INTERVENTIONS:
Biological: Autologous Concentrated Plasma — Autologous blood products have created a growing interest for use in a number of orthopedic therapies. The healing effects of plasma are supported by growth factors released by platelets. These growth factors induce a healing process wherever they are applied. The Arthrex ACP System is a cost-effective method of concentrating growth factors for therapeutic use.
  Other Names: ACP
  Arms: Fusion + ACP +DBM; Fusion+ACP+Autograft

SUMMARY:
To compare the outcomes of patients who undergo three different types of surgeries for ankle fusion and reconstruction.

DETAILED DESCRIPTION:
It is understood that an elevated concentration of platelets in the mix of the arthrodesis construct applied intra-operatively to the bony surface, has osteo-generating and enhanced wound healing properties. With that knowledge there is a clinical need and enthusiasm for the application of concentrated platelets, which release a large quantity of growth factors to encourage recovery in non healing injuries or surgical sites. This study represents an effort to more clearly define the true clinical outcomes with or without biologic enhancement, and fulfills a need for fortifying evidence concerning the efficacy of ACP in live human bone healing-- based on radiographic and CT scans.

ELIGIBILITY:
Inclusion Criteria:

* patients whom present the need for the elective surgery

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Shurnas, Principal Investigator — Columbia Orthopaedic Group
Locations (1):
- Columbia Orthopedic Group, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fusion+ACP+Autograft: Standard anatomic reduction will be adhered to- neutral alignment will be employed (5° valgus, external rotation and neutral foot dorsiflexion). The arthrodesis undertaken for all will be the standard arthroscopic ankle arthrodesis with portals to the ankle (anterior medial / anterior lateral), skin incision only technique with dissection through the capsule and penetration to the joint. Standard debridement of the gutters, tibia osteophyte, tibia-talor joint resection and autograft preparation will be performed in the joint. Depending on randomization of the subject, (Autologous concentrated Plasma)ACP-A or ACP-DBM mixture will be added to the arthrodesis site with the joint taken through range of direct motion and reduced.
  Autologous Concentrated Plasma: Autologous blood products have created a growing interest for use in a number of orthopedic therapies. The healing effects of plasma are supported by growth factors released by platelets. These growth factors induce a h
Period: Overall Study
Arm/Group | Fusion+ACP+Autograft | Fusion + ACP +DBM | Standard-Fusion +Autograft Only
Started | 6 | 4 | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 4 | 0
Not completed — Death of PI | 6 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fusion+ACP+Autograft: Standard anatomic reduction will be adhered to- neutral alignment will be employed (5° valgus, external rotation and neutral foot dorsiflexion). The arthrodesis undertaken for all groups will be the standard arthroscopic ankle arthrodesis with portals to the ankle (anterior medial / anterior lateral), skin incision only technique with dissection through the capsule and penetration to the joint. Standard debridement of the gutters, tibia osteophyte, tibia-talor joint resection and autograft preparation will be performed in the joint. Depending on randomization of the subject, (Autologous concentrated Plasma)ACP-A or ACP-DBM mixture will be added to the arthrodesis site with the joint taken through range of direct motion and reduced.
  Autologous Concentrated Plasma: Autologous blood products have created a growing interest for use in a number of orthopedic therapies. The healing effects of plasma are supported by growth factors released by platelets. These growth factors induce a h
- Total: Total of all reporting groups
Arm/Group | Fusion+ACP+Autograft | Fusion + ACP +DBM | Standard-Fusion +Autograft Only | Total
Number analyzed (Participants) | 6 | 4 | 0 | 10
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 2 | 4 |  | 6
  >=65 years | 4 | 0 |  | 4
Gender [Number; unit: participants]
  Female | 3 | 4 |  | 7
  Male | 3 | 0 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: CT Scan for Fusion Analysis
Description: There will be no outcome analysis for the CT scan performed on the 10 patients due to the death of the primary investigator.
Time Frame: 8 weeks post op.
Arm/Group | Fusion+ACP+Autograft | Fusion + ACP +DBM | Standard-Fusion +Autograft Only
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Fusion+ACP+Autograft | Fusion + ACP +DBM | Standard-Fusion +Autograft Only
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No